CLINICAL TRIAL: NCT06314711
Title: Tumor Volume and Margin Assessment with Ex Vivo 3D-ultrasound After Transoral Robotic Surgery for Oropharyngeal Squamous Cell Carcinoma
Brief Title: Ex Vivo 3D-ultrasound for Oropharyngeal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin Garset-Zamani, MD, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ex Vivo US for OPC
Record Dates: First submitted 2024-03-06; First posted 2024-03-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Post-operative ex vivo 3D ultrasound (Experimental): 3D ultrasound of surgical specimen
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — High-frequency ultrasound of ex vivo specimen

SUMMARY:
Patients with biopsy-verified oropharyngeal squamous cell carcinomas treated with transoral robotic surgery are included. Immediately post-operatively, freshly resected specimens are examined with ex vivo 3D ultrasound (US).

Ex vivo 3D US will be used to match US slices of the specimen with corresponding histopathology slices. The US slices will be reviewed by a panel of head and neck surgeons blinded to histopathology.

The primary aim is to explore perioperative ex vivo 3D US for oropharyngeal tumor detection, delineation from normal tissue, tumor size and volume, and margin assessment.

DETAILED DESCRIPTION:
The purpose of the study is to determine the accuracy of ex vivo 3D ultrasound (US) for detecting and delineating tumor tissue of the tonsils and base of tongue post-operatively. This is a quick technique that may provide valuable information for the surgeon that can potentially improve treatment outcomes.

Placing the surgical specimen in a water bath allows for an US swipe to be performed without compressing the specimen. This reduces the deformation of the specimen by removing the pressure from conventional US scanning. A video clip can be captured by swiping across the specimen in the water bath. By motorizing this motion, the video can be converted into a 3D volume due to the known number of video frames and a constant swiping speed.

We will correlate the ex vivo 3D US scans to histopathology for the following analyses:

* Four surgeons blinded to histopathology will rate each included case in terms of tumor visibility on ex vivo 3D US scans. If visible, the surgeons will mark the tumor and the healthy tissue.
* Tumor and margins will be correlated to histopathology pre- and post-formalin fixation on a subset of cases to explore the proportion of tissue shrinkage from formalin fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patients surgically treated with transoral robotic surgery for oropharyngeal squamous cell carcinoma.

Exclusion Criteria:

* Patients from the QOLATI trial (NCT04124198)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Blind-assessed tumor size from fresh ex vivo US | day 1
  Tumor width and thickness (mm) estimated by blinded perioperative ex vivo 3D-US
Blind-assessed deep and lateral margin measurements on fresh ex vivo US | day 1
  Deep and lateral margin measurements (mm) by blinded perioperative ex vivo 3D-US.

SECONDARY OUTCOMES:
Fresh vs formalin-fixed ex vivo US tumor volume | day 1
  Comparison of tumor volumes (mm^3) estimated by ex vivo perioperative 3D-US before and after formalin fixation.
Margin involvement (categorical) | day 1
  Blinded evaluation of involved tumor margins (involved vs not involved)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Otorhinolaryngology, Head & Neck Surg, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makouei F, Agander TK, Ewertsen C, Sondergaard Svendsen MB, Norling R, Kaltoft M, Hansen AE, Rasmussen JH, Wessel I, Todsen T. 3D Ultrasound and MRI in Assessing Resection Margins during Tongue Cancer Surgery: A Research Protocol for a Clinical Diagnostic Accuracy Study. J Imaging. 2023 Aug 28;9(9):174. doi: 10.3390/jimaging9090174. PMID 37754938